CLINICAL TRIAL: NCT00488176
Title: Comparison of the Effect of Montelukast and Cetirizine on Allergic Inflammation Measured by Exhaled Nitric Oxide Concentration in Children With Seasonal Allergic Rhinitis
Brief Title: Comparison of the Effect of Montelukast and Cetirizine on Allergic Inflammation in Children With Allergic Rhinitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN/94/07KE
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: seasonal allergic rhinitis; children; montelukast; cetirizine
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): monteluksat sodium
  Interventions: Drug: montelukast
- 2 (Active Comparator): cetirizine
  Interventions: Drug: cetirizine
- 3 (Active Comparator): montelukast sodium and cetirizine
  Interventions: Drug: montelukast and cetirizine
- 4 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast — montelukast sodium
  Other Names: montelukast sodium
  Arms: 1
Drug: cetirizine — cetirizine
  Arms: 2
Drug: montelukast and cetirizine — montelukast and cetirizine
  Arms: 3
Drug: placebo — placebo
  Arms: 4

SUMMARY:
The aim of this study is to compare the effect of montelukast and cetirizine on allergic inflammation measured by exhaled nitric oxide concentration in children with seasonal allergic rhinitis.

DETAILED DESCRIPTION:
During the pollen season children with seasonal allergic rhinitis without concomitant asthma are at risk of having allergic inflammation in the lower respiratory tract. About 60% of children with seasonal allergic rhinitis present bronchial hyperresponsiveness and signs and symptoms of asthma.

The aim of this study is to compare the effect of montelukast and cetirizine on allergic inflammation measured by exhaled nitric oxide concentration in children with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms of seasonal allergic rhinitis during last two seasons, moderate and severe according to ARIA guidelines

Exclusion Criteria:

* diagnosis of bronchial asthma
* allergy to perennial allergens
* specific immunotherapy
* other chronic diseases
* tobacco smoking
* acute respiratory tract infection
* excluded drugs: inhaled and systemic glucocorticosteroids

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2007-04; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
exhaled nitric oxide concentration | baseline (first visit), after 4 weeks (second visit) and after 6 weeks from second visit (third visit)

SECONDARY OUTCOMES:
symptoms score (based on PAQLQ), bronchial hyperresponsiveness with methacholine, spirometry, PEFR measurements | baseline (first visit), after 4 weeks (second visit) and after 6 weeks from second visit (third visit)

CONTACTS AND LOCATIONS:
Overall Officials: Violetta Ścibiorek, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD PhD Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz Lodz, Poland, Lodz, Poland